CLINICAL TRIAL: NCT03952078
Title: A Phase 1/1b Dose-Escalation Trial Evaluating CPI-818, an Oral Interleukin-2-Inducible T-Cell Kinase Inhibitor, in Subjects With Relapsed/Refractory T-Cell Lymphoma
Brief Title: A Dose Escalation Study Evaluating CPI-818 in Relapsed/Refractory T-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Corvus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPI-818-001
Record Dates: First submitted 2019-05-07; First posted 2019-05-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: T-cell Lymphoma
Keywords: CTCL; PTCL
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CPI-818 Dose Escalation (Experimental): Participants will receive CPI-818 capsule, orally, twice per day at an assigned dose, till disease progression, complete response or remission (CR) for >2 months or if dose determined to be unsafe.
  Interventions: Drug: CPI-818
- CPI-818 Dose Expansion phase (Experimental): Participants with different T-cell lymphoma sub-types will receive CPI-818 capsules at the specific dose selected from the Dose escalation phase of the study.
  CPI-818 capsules at the selected dose will be taken orally, twice per day until disease progression or CR for > 2 months.
  Interventions: Drug: CPI-818

INTERVENTIONS:
Drug: CPI-818 — Interleukin-2 inducible T-cell Kinase Inhibitor

SUMMARY:
This is a Phase 1/1b, open-label, first in human study of CPI-818, an oral interleukin-2-inducible tyrosine kinase (ITK) inhibitor for the treatment of relapsed/refractory (R/R) T-cell lymphoma.. This trial will study the safety, tolerability, and anti-tumor activity of CPI-818 as a single drug.

DETAILED DESCRIPTION:
This is a Phase 1/1b, open-label, first in human study of CPI-818, an oral interleukin-2-inducible tyrosine kinase (ITK) inhibitor for the treatment of relapsed/refractory (R/R) T-cell lymphoma.. This trial will study the safety, tolerability, and anti-tumor activity of CPI-818 as a single drug. This trial is composed of dose escalation and dose expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Histologically confirmed evidence of T-cell lymphoma
* Measurable disease.
* Adequate organ function.
* At least 2 standard therapies for advanced or recurrent disease or had a disease for which there is no more than one established therapy.

Exclusion Criteria:

* Treatment with systemic immunosuppressive medication.
* History of allogeneic hematopoietic stem cell transplantation.
* History of primary immunodeficiency, solid organ transplantation.
* History of opportunistic infection within 180 days of starting study drug.
* Females who are pregnant, lactating, or intend to become pregnant
* History of invasive prior malignancy that required systemic therapy within last 3 years.
* Concomitant use of strong inhibitors or inducers of CYP3A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Estimated)
Dates: Start 2019-05-03 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events following treatment with CPI 818 to establish the safety and tolerability with increasing dose | First dose until 30 days after treatment stop
Incidence and nature of dose limiting toxicities (DLTs) of CPI 818 to establish either the maximum tolerated dose (MTD) or the maximum administered dose (MAD) of CPI 818 | Up to approximately 21 days after first dose

SECONDARY OUTCOMES:
Area under the curve (AUC) of CPI-818 in blood samples to evaluate the pharmacokinetic profile of CPI 818 | Day 1, 2, 8, 15 of Cycle 1, Day 1 and 2 of Cycle 3, and Day 1 for all even number Cycles. Each Cycle is 21 days.
Maximum serum concentration (Cmax) of CPI-818 in blood samples to evaluate the pharmacokinetic profile of CPI 818 | Day 1, 2, 8, 15 of Cycle 1, Day 1 and 2 of Cycle 3, and Day 1 for all even number Cycles. Each Cycle is 21 days.
Objective response rate per Laguno Classification for CTCL and Consensus Statement for Response for CTCL to assess the anti-tumor activity of CPI 818 in subjects with R/R T cell lymphoma | From start of treatment through end of study treatment, up to approximately 24 months
Evaluate total percentage of tumor gene expression in post-treatment blood and tumor samples to evaluate pharmacodynamic changes with treatment. | Day 1, 2, 8, 15 of Cycle 1, Day 1 and 2 of Cycle 3, and Day 1 for all even number Cycles. Each Cycle is 21 days.
Evaluate overall percentage of malignant cells in post-treatment blood and tumor samples to evaluate pharmacodynamic changes with treatment. | Day 1, 2, 8, 15 of Cycle 1, Day 1 and 2 of Cycle 3, and Day 1 for all even number Cycles. Each Cycle is 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Mahabhashyam, MD, MPH, Study Director — Corvus Pharmaceuticals
Locations (22):
- United States (6):
  - Stanford University, Palo Alto, California
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Australia (4):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Epworth Healthcare, Melbourne, Victoria
- China (5):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Boren Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Shanghai East Hospital, Pudong, Shanghai Municipality
  - Henan Cancer Hospital, Henan, Zhengzhou
- South Korea (7):
  - Seoul National University Hospital, Seoul, Gyeonggido
  - Asan Medical Center, Seoul, Gyeonggido
  - Samsung Medical Center, Seoul, Gyeonggido
  - Seoul St. Mary's Hospital, Seoul, Gyeonggido
  - Inje University Busan-Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Gachon University, Incheon